CLINICAL TRIAL: NCT07123805
Title: ACU_Knee - Role of Acupuncture in Knee Prosthetic Surgery: Analgesia, Functional Outcome and Inflammatory Markers
Brief Title: ACU_Knee: Role of Acupuncture in Knee Prosthetic Surgery
Acronym: ACU_Knee
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Debora Passador, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACU_Knee
Record Dates: First submitted 2025-03-12; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-02

CONDITIONS: Acupuncture Analgesia; Acupuncture; Acupuncture Therapy; Total Knee Anthroplasty; Postoperative Pain Management; Pain Threshold; Shoulder Pain; Laparoscopies; Acupuncture Ear
Keywords: acupuncture; total knee arthroplasty; pain
MeSH Terms: conditions — Shoulder Pain; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard group (No Intervention): the anesthesiological treatment will be the one routinely used at our UOC: mild sedation with midazolam 1-2mg ev LRA subarachnoid with Levobupivacaine 0.5% 10-12mg tranexamic acid 1g ev. dexamethasone 4mg ev pre-operative analgesic block of the saphenous nerve with L-bupivacaine 0.5% 15ml, ultrasound-guided technique: pre-operative iPACK Block (Interspace between the Popliteal Artery and Capsule of the Knee) with L-bupivacaine 0.375% 20ml, ultrasound-guided technique; intraoperative analgesic therapy: Ketorolac 15mg + Paracetamol 1000mg ev post-operative analgesic therapy: paracetamol 1000mg ev every 8 hours; ibuprofen 400mg cp every 8 hours; tapentadol 50mg cp every 12 hours; rescue therapy (to be administered in case of NRS > 4): Oxycodone + Paracetamol 5/325mg, 1cp every 30 minutes, for a maximum of 4cp/day.
- Acupuncture group (Active Comparator): In the Acu group, acupuncture and auriculotherapy will be added to the standard treatment: patients will undergo three/four sessions of manual acupuncture lasting 20 minutes, the first in the immediate pre-operative period and the subsequent ones at a distance of 24, 48, 72 hours from surgery. The treatment includes manual acupuncture applied to specific points: LI4, LV3 and ST36 bilaterally and monolaterally SP6 and GB34, ipsilateral to the knee to be prostheticized. Furthermore, auricolar needles will be positioned, before surgery, for self-stimulation of the auriculotherapy points corresponding to Shen Men bilaterally and the knee point ipsilateral to the surgical side.
  Interventions: Device: Acupuncture group

INTERVENTIONS:
Device: Acupuncture group — In the Acu group, acupuncture and auriculotherapy will be added to the standard treatment: patients will undergo three/four sessions of manual acupuncture lasting 20 minutes, the first in the immediate pre-operative period and the subsequent ones at a distance of 24, 48, 72 hours from surgery. The treatment includes manual acupuncture applied to specific points: LI4, LV3 and ST36 bilaterally and monolaterally SP6 and GB34, ipsilateral to the knee to be prostheticized. Furthermore, auricolar needles will be positioned, before surgery, for self-stimulation of the auriculotherapy points corresponding to Shen Men bilaterally and the knee point ipsilateral to the surgical side.
  Arms: Acupuncture group

SUMMARY:
Post-operative analgesia after total knee arthroplasty (TKA) has always been a challenge in the anesthesiological setting, having to combine good pain control and the need for early mobilization, both factors that can affect the quality of rehabilitation treatment, prosthetic functional outcome, the onset of chronic pain, joint stiffness and the consequent quality of life of the patient. Recent loco-regional anesthesia (LRA) techniques have made an essential contribution to peri-operative management in the fast-track perspective of surgery, in terms of optimization of analgesia and rapid functional recovery. Inadequate post-operative analgesia, by affecting the normal rehabilitation pathway, is associated with medium-long term complications, such as chronic pain, joint stiffness and patient dissatisfaction, which often compromise functional autonomy and quality of life of the patient and may require invasive treatments (surgical revision, unlocking under general anesthesia). The local and systemic inflammatory state, evidenced by peri-operative dosage of specific biomarkers, appears to be related to prosthetic outcome.

DETAILED DESCRIPTION:
Objectives, "The purpose of the study is to evaluate whether acupuncture, a technique recognized in the literature for its analgesic, anti-inflammatory and immunomodulatory effect, can affect: acute pain control and chronic pain prevention, functional outcome and subjective patient satisfaction. In particular, the investigators propose to define, through clinical evaluation and blood dosage of inflammation mediators, the anti-inflammatory effect of acupuncture, whether this affects the trend of inflammatory biomarkers and whether it can influence the functional result and the establishment of post-operative joint stiffness. Primary endpoint: to evaluate the efficacy of acupuncture on post-operative pain control at 36-48 hours after surgery, when moderate-severe pain occurs, due to the resolution of peripheral blocks. This role will be evaluated in relation to: total opioid consumption and the onset of side effects (nausea/vomiting, constipation, sedation), time out-of-bed and effect on the rehabilitation pathway, patient satisfaction. The medium/long-term functional outcome will be analyzed at one, three, six and twelve months after surgery. Secondary endpoint: to evaluate the effect of acupuncture on the modulation of systemic inflammatory response through the analysis of specific serum biomarkers and to evaluate their correlation with functional outcome and the onset of chronic pain." Inclusion/exclusion criteria Inclusion criteria: patients undergoing total knee replacement for primary osteoarthritic degeneration, elective monolateral surgery, patients capable of informed consent.

Exclusion criteria: age < 18 years, total knee replacement for causes other than primary osteoarthritis (e.g. post-traumatic arthritis), revision surgery, contraindications to loco-regional anesthesia, contraindications to therapy with NSAIDs, cortisones and paracetamol, chronic assumption of opiates, use of corticosteroids in the six months prior to surgery, periarticular infiltration in the three months prior to surgery, patients with rheumatoid arthritis or autoimmune disorders, patients on therapy with biological drugs, ASA class > 3, pregnant women, active infection in antibiotic treatment.

Methods: Patients candidates for elective, monolateral, total knee replacement will be enrolled. The following data will be collected: demographic characteristics; comorbidities and psychological status (SF-12 score); pre-operative severity score (WOMAC Score); pre-operative pain assessment (NRS scale). For all patients, the anesthesiological treatment will be the one routinely used in the investigators' UOC : mild sedation with midazolam 1-2mg ev LRA subarachnoid with Levobupivacaine 0.5% 10-12mg tranexamic acid 1g ev. dexamethasone 4mg ev pre-operative analgesic block of the saphenous nerve with L-bupivacaine 0.5% 15ml, ultrasound-guided technique: pre-operative iPACK Block (Interspace between the Popliteal Artery and Capsule of the Knee) with L-bupivacaine 0.375% 20ml, ultrasound-guided technique; intraoperative analgesic therapy: Ketorolac 15mg + Paracetamol 1000mg ev post-operative analgesic therapy: paracetamol 1000mg ev every 8 hours; ibuprofen 400mg cp every 8 hours; tapentadol 50mg cp every 12 hours; rescue therapy (to be administered in case of NRS > 4): Oxycodone + Paracetamol 5/325mg, 1cp every 30 minutes, for a maximum of 4cp/day. Patients will be divided into two groups: Acu vs Standard. In the Standard group, the treatment will be the one described above. In the Acu group, acupuncture and auriculotherapy will be added to the standard treatment: patients will undergo three/four sessions of manual acupuncture lasting 20 minutes, the first in the immediate pre-operative period and the subsequent ones at a distance of 24, 48, 72 hours from surgery. The treatment includes manual acupuncture applied to specific points: LI4, LV3 and ST36 bilaterally and monolaterally SP6 and GB34, ipsilateral to the knee to be prostheticized. Furthermore, auricolar needles will be positioned, before surgery, for self-stimulation of the auriculotherapy points corresponding to Shen Men bilaterally and the knee point ipsilateral to the surgical side. The patient will be instructed on how to self-stimulate these auricular points during hospitalization. Patients will be evaluated at 24, 48, 72, 96 hours after surgery; post-operative parameters: evaluation of dynamic and resting pain (NRS scale), assumption of rescue analgesics; trend of vital parameters (HR, NIBP, RR, SpO2); incidence of adverse events and complications; functional outcomes: post-operative joint mobility parameters (ROM, Range of Motion, active and passive), time out-of-bed, resumption of ambulation, length of hospital stay (surgery-end of rehabilitation); patient-reported outcomes and related measures: Patient-Reported Outcome Measures (PROMs) and, specifically, Knee Injury and Osteoarthritis Outcome Score (KOOS); satisfaction questionnaire. In addition to biomarkers such as CRP and N/L ratio, routinely measured in the post-operative period, blood dosages of specific inflammation mediators (IL2 IL6 IL8 IL10 IFNy TNFa) will be performed in three moments: pre-operative, 48 hours and one month after surgery. The medium/long-term re-evaluation of enrolled patients will coincide with the outpatient checks normally prescribed, at a distance of one, three, six and twelve months post-TKA, and will include: evaluation of dynamic and resting pain (NRS scale); need for analgesic assumption; post-operative joint mobility parameters (ROM, Range of Motion, active and passive), patient-reported outcomes and related measures: Patient-Reported Outcome Measures (PROMs) and, specifically, Knee Injury and Osteoarthritis Outcome Score (KOOS); satisfaction questionnaire. In case the patient is unable to go to UOC for the checks scheduled after three months from surgery, the evaluation will take place by telephone.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18 years
* Patients capable of providing informed consent
* Unilateral total knee replacement surgery
* Indication for surgery: primary osteoarthritis degeneration
* Surgery performed electively

Exclusion Criteria:

* Patients aged < 18 years
* Patients incapable of providing informed consent
* Patients with ASA class > 3
* Pregnant women
* Patients with rheumatoid arthritis or other autoimmune disorders
* Patients with active infection under antibiotic treatment
* Patients on chronic opioid therapy
* Patients on chronic biological drug therapy
* Patients with a history of corticosteroid use in the six months prior to surgery
* Patients with a history of periarticular infiltration in the three months prior to surgery
* Patients in whom loco-regional anesthesia is contraindicated
* Patients in whom NSAID, cortisone, and paracetamol therapy is contraindicated
* Bilateral total knee replacement surgery or prosthetic revision surgeries
* Indication for surgery for causes other than primary osteoarthritis degeneration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Quantity of opioid rescue medication taken by the patient | 48-96 hours
  Number of tablets taken daily and overall between 48 and 96 hours post-surgery

SECONDARY OUTCOMES:
Time to first dose | one, three, six, and twelve months
  Time between surgery and the first dose of rescue opioid

OTHER OUTCOMES:
Appearance of side effects related to opioid use during the first 96 hours of hospitalization | One, three, six, and twelve months
  Safety in terms of local tolerability in patients in the acupuncture treatment arm and systemic adverse events
Pain perceived by the patient according to the NRS pain assessment scale at rest and dynamic | One, three, six, and twelve months
Patient's sleep quality | One, three, six, and twelve months
  Analysis of the relaxing effect and modulation on sleep quality during the first 96 hours of hospitalization using the Richards-Campbell Sleep Questionnaire
Time out-of-bed | One, three, six, and twelve months
  The variation in the time interval between surgery and the resumption of standing
The overall effect on the rehabilitation path | One, three, six, and twelve months
  Assessing the range of joint motion during active and passive physical therapy, and the resumption of independent walking
Time to resume walking | One, three, six, and twelve months
Analysis of Knee Injury and Osteoarthritis Outcome Score (KOOS) | One, three, six, and twelve months
Analysis of the International Knee Documentation Committee (IKDC) Subjective Knee Form | One, three, six, and twelve months
The potential effect of acupuncture on modulating the systemic inflammatory response | 48 hours and one month
  Blood dosage of specific inflammatory mediators

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo - SC AR3 - Anestesia e Terapia Intensiva Postchirurgica, Pavia, Pavia, Italy